CLINICAL TRIAL: NCT04857086
Title: A Multi-center Study to Observe Five-year Outcomes of the Initial Management in Patients With Differentiated Thyroid Cancer in the Real World in China (The Second Stage of DTCC)
Brief Title: The Initial Management in Patients With Differentiated Thyroid Cancer in the Real World in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); West China Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Sir Run Run Shaw Hospital (Other); China-Japan Union Hospital, Jilin University (Other); Chinese PLA General Hospital (Other); Tongji Hospital (Other); First Hospital of China Medical University (Other); Gansu Cancer Hospital (Other)
Responsible Party: Principal Investigator, Tao Huang, Director of breast and thyroid department of Wuhan Union Hospital，Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: MS200007_0003
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Differentiated Thyroid Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group1: About 1400 DTC patients with more than 5 years long-term follow-up from the date of signing the informed consent form (ICF) in DTCC 1st to signing ICF in DTCC 2nd will be collected data retrospectively.

SUMMARY:
* To find out the gap between real-world clinical practice and guideline recommendations in initial management of DTC patients
* To observe the characteristics of patients who achieved and did not achieve TSH target value after five year follow-up
* To assess response to initial therapy in patients who undergo total or neartotal thyroidectomy and RAI remnant ablation after five year follow-up (according to an modified dynamic risk stratification system)
* To observe the recurrence status after five year follow-up

DETAILED DESCRIPTION:
The DTCC 2nd will follow DTCC 1st and observe the long-term efficacy of initial management including surgery treatment, 131I therapy and TSH suppression therapy. It will involve nine hospitals which have participated in the first stage, and continually to observe the DTC patients who were recruited. The patients with more than 5 years long-term follow-up from the date of signing the informed consent form (ICF) in DTCC 1st to signing ICF in DTCC 2nd will be collected data retrospectively. For those follow-up less than 5 years, in addition to the retrospective data collection, one prospective visit will be conducted.

Primary endpoint(s)

1.Five-year accumulated recurrence rate

Secondary endpoint(s)

1. Disease-free survival (DFS)
2. Overall survival (OS)
3. Response to therapy
4. Re-operation rate
5. Time weighted TSH level (TW-TSH)
6. Adverse events related to L-T4 therapy (ADRs)
7. Median follow-up years

ELIGIBILITY:
Inclusion Criteria:

- Patients who had been recruited into DTCC 1st study will be enrolled.

Exclusion Criteria:

* Other malignant tumors;

  * Severe organ damage such as heart failure of New York Heart Association classes III-IV, liver failure, respiratory failure, renal failure, etc.;

    * Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent; ④ Legal incapacity or limited legal capacity; ⑤ Unwilling to be followed up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients are those who had been recruited into the first stage of DTCC study, including intermediate and high risk DTC patients.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-03-28 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | five year
  Five-year accumulated recurrence rate

SECONDARY OUTCOMES:
Disease-free survival (DFS) | five year
  Evaluated from the date of first-time thyroidectomy to the first to the progression date or death related to disease progression, whichever occurs first
Overall survival (OS) | five year
  Evaluated from the date of first-time thyroidectomy to the death for any reason
Response to therapy | five year
  Presented by number of patients and proportions
Re-operation rate | five year
  the percentage of patients accepting operation due to DTC progression.
Time weighted TSH level (TW-TSH) | five year
  Calculated by specific formula
Adverse events related to L-T4 therapy (ADRs) | five year
  The number of patients, number of ADRs and the incidence rate will be summarized for L-T4 therapy
Median follow-up years | five year
  Gained by statistical summary of median follow-up time

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Not yet